CLINICAL TRIAL: NCT01306773
Title: Convalescent Plasma Treatment in Patients With Severe 2009 H1N1 Infection: a Prospective Cohort Study
Brief Title: Convalescent Plasma Treatment in Severe 2009 H1N1 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Dr Ivan FN Hung, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKU-CP1
Record Dates: First submitted 2011-01-05; First posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-03

CONDITIONS: Influenza A
Keywords: Influenza A; convalescent plasma; death
MeSH Terms: conditions — Death | interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- H1N1 convalescent plasma and oseltamivir (Active Comparator): Oseltamivir 75mg bid orally during ICU hospitalization + 500mL convalescent plasma
  Interventions: Drug: H1N1 convalescent plasma and oseltamivir
- Oral Oseltamivir alone (Active Comparator): Oseltamivir 75mg bid during ICU hospitalization
  Interventions: Drug: Oral Oseltamivir alone

INTERVENTIONS:
Drug: H1N1 convalescent plasma and oseltamivir — Oseltamivir 75mg bid orally during ICU hospitalization + 500mL convalescent plasma containing >= 1:160 of neutralizing antibody to Pandemic influenza A H1N1
  Arms: H1N1 convalescent plasma and oseltamivir
Drug: Oral Oseltamivir alone — Oral Oseltamivir 75mg bid during ICU hospitalization
  Arms: Oral Oseltamivir alone

SUMMARY:
Treatment of severe 2009 H1N1 infection with convalescent plasma will reduce mortality.

DETAILED DESCRIPTION:
Patients presented with severe 2009 H1N1 infection responded poorly to antiviral agents. Meta-analysis of reports from 1918 H1N1 pandemic suggested that convalescent plasma might be an effective treatment option for patients with severe 2009 H1N1 infection.

ELIGIBILITY:
Inclusion Criteria:

* adult patients ≥ 18 years old with written informed consent given by patient or next-of-kin
* laboratory confirmatory diagnosis of 2009 H1N1 infection by positive RT-PCR from respiratory specimens
* required intensive care within 7 days of onset of symptoms

Exclusion Criteria:

* age 18 years old or below
* known hypersensitivity to immune globulin
* known IgA deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Death | Participants are followed until death or discharge from ICU (average 2 weeks)
  mortality during hospitalization directly related to H1N1 2009 infection

SECONDARY OUTCOMES:
Complication | Participants are followed until death or discharge from ICU (average 2 weeks)
  including pneumonia, ARDS, renal failure, heart failure and secondary infection
Length of stay in ICU | Participants are followed until death or discharge from ICU (average 2 weeks)
  days of stay in ICU
Adverse events secondary to the convalescent plasma treatment | Participants are followed until death or discharge from ICU (average 2 weeks)
  Allergic reaction (including anaphylaxis), acute renal failure, fluid overload
Time on respiratory support | Participants are followed until death or discharge from ICU (average 2 weeks)
  including ventilator, CPAP and BiPAP
Change in viral load | Participants are followed until death or discharge from ICU (average 2 weeks)
  Daily measurement of H1N1 2009 viral load
Change in cytokine level | Participants are followed until death or discharge from ICU (average 2 weeks)
  daily measurement of cytokine level (serum)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN HUNG, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong SAR, China